CLINICAL TRIAL: NCT06631534
Title: Effect of Dexmedetomidine Supplementation to General Anaesthesia in Paediatric Transcatheter Closure of Atrial Septal Defect
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Adel Okasha, Assistant Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0201930
Record Dates: First submitted 2024-09-25; First posted 2024-10-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Atrial Septal Defect (ASD); Dexmedetomidine; Delirium - Postoperative; Stress Response
Keywords: Atrial septal Defect; ASD; Dexmedetomidine; Echocardiography; Cardiac index; PAED; VTI; Norepinephrine; Corisol
MeSH Terms: conditions — Heart Septal Defects, Atrial; Emergence Delirium; Fractures, Stress | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group GD (Active Comparator): Anesthesia induction and maintenance with sevoflurane inhalational anesthesia in addition dexmedetomidine diluted in normal saline (NS) to a concentration of 4ug/ml (in a 50 ml syringe) bolus dose will be administered through the IV catheter at 1 ug/kg over 10 minutes, followed by an infusion rate of dexmedetomidine 0.5ug/kg/hr with use of a syringe pump.
  Interventions: Drug: Dexmedetomidine
- Group GS (Placebo Comparator): Anaesthesia induction and maintenance with sevoflurane inhalational anaesthesia in addition a 50 ml syringe admisinstered at the same initial rate and maintenance rate as would a vloume-matched dexmedetomidine syringe. Syringes will be prepared by an independent party.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 1ug/kg bolus administered over 10 minutes followed by a continuous infusion of 0.5ug/kg/hr
  Arms: Group GD
Drug: Saline (NaCl 0,9 %) (placebo) — Saline (placebo)
  Arms: Group GS

SUMMARY:
The aim of this randomized trial is to determine efficacy of dexmedetomidine in improving quality of recovery in pediatric patients undergoing interventional catheter closure of ASD while maintaining the hemodynamic parameters. Additionally he stress reducing effects of dexmedetomidine will be investigated in this population .

The main questions it aims to answer are:

Does Dexmedetomidine maintain stable hemodynamics in pediatric patients undergoing transcatheter ASD Closure while improving their quality of recovery?

Does dexmedetomidine prolong duration of recovery and time to extubation in pediatric patients ?

Does dexmedetomidine exert stress reducing properties in this population?

Participants will:

Either be administered Dexmedetomidine in a loading/maintenance regimen or a placebo, with hemodynamics being monitored at the baseline, intraoperatively and postoperatively, with recovery time and quality of recovery especially emergence delirium being monitored. Stress hormone levels will be sampled at baseline and postoperatively.

DETAILED DESCRIPTION:
Atrial Septal Defect (ASD) is one of the most common congenital anomalies in pediatric and even in adult population, it is associated with a left-to-right shunt resulting in right ventricular (RV) volume overload and increase in pulmonary blood flow eventually culmination in right ventricular heart failure (RVHF) and pulmonary hypertension.

Percutaneous closure of ASD was devised nearly a half century ago, and now constitutes a viable alternative to the standard approach of surgical closure. Anesthesia for pediatric patients undergoing percutaneous closure involves a spectrum from sedation to general anesthesia using a variety of drugs according to institutional protocol.

Stress response represents the sum of metabolic nd hormonal perturbations initiated by the hypothalamo-pituitary-adrenal axis in response to the surgical stimulus.

Dexmedetomidine is an α2-adrenoreceptor agonist possessing stress ameliorating effects exerted on the central sympathetic outflow. It can be used either alone in sedation or as supplementation to general anesthesia. It possesses a remarkable hemodynamic stability profile and due to its prolonged duration of action, it plays a significant role in reducing emergence delirium.

This study aims at evaluating utility of dexmedetomidine as a supplementary agent to general anesthesia on hemodynamic stability / cardiac output, reduction of pediatric emergence delirium and stress hormone levels in pediatric patients undergoing transcatheter closure of ASD.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients 3-12 years of age admitted for device closure of ASD secundum

Exclusion Criteria:

* ASA IV, V
* Neurological problems (cerebral palsy, mental retardation, etc.,)
* Children with chromosomal abnormalities or other multiple congenital anomalies or other complex cardiac anomalies
* Hepatic or renal insufficiency
* History of allergy to the drugs used
* Previous Cardiac Surgery

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Parameters - Cardiac Output | Baseline , Perioperatively
  Cardiac Output/Cardiac index assessed via VTI derived Stroke volume
Hemodynamic Parameters - Heart Rate | Baseline , Perioperatively
Hemodynamic Parameters - Mean Arterial Blood Pressure | Baseline , Perioperatively

SECONDARY OUTCOMES:
Quality of Recovery | Perioperatively
  Quality of recovery will be assessed in paediatric ICU using the paediatric anaesthesia emergence delirium (PAED) scores every 5 minutes after awakening for 30 minutes
G. Recovery Time | Perioperatively
  The time from application of groin bandage to reach a modified Steward score of ≥ 6
Time to extubation | Perioperatively
  Time from applying of groin bandage and cessation of anaesthetic, to removal of ETT
Stress Hormones | Baseline , Perioperatively
  Norepinephrine level
Stress Hormones | Baseline , Perioperatively
  Cortisol Level
Side Effects | Perioperatively
  Clinically significant Bradycardia: HR less than 60 or decrease 30% Clinically significant Tachycardia: HR increase 30% Clinically significant Hypotension: MAP decrease 30% Clinically significant Hypertension: MAP increase 30% Nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Hospitals - Semouha, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No